CLINICAL TRIAL: NCT05002322
Title: Scaling Out and Scaling Up the Systems Analysis and Improvement Approach to Optimize the Hypertension Diagnosis and Care Cascade for HIV-infected Individuals
Brief Title: Expanding Health Systems Research to Optimize Hypertension Care Cascade in HIV-Infected Individuals in Mozambique
Acronym: SCALESAIAHTN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eduardo Mondlane University (Other)
Collaborators: University of Washington (Other); Instituto Nacional de Saúde, Mozambique (Other Government); Mozambique Institute for Health Education and Research (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: SCALESAIA2020; 4UH3HL156390-03 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-08-12 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: Systems analysis and improvement approach (SAIA),; Hypertension; CFIR; ORIC; Process mapping; Cascade analysis; Continuous quality improvement; Implementation science; Systems engineering; HIV
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: phased-in (stepped wedge) design with random assignment of two districts to each of the three nine-month intervention waves, to reach six districts in Maputo Province by the end of the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention health facilities (Experimental): Health facilities implement the optimization of the cascade under research team support and continuous supervision.
  Interventions: Other: Systems Analysis and Improvement Approach
- Control (No Intervention): Health facilities prior to intensive phase receive standard supervision without research team support

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach — Intensive phase: district MOH supervisors receive a one-week training on SAIA-HTN. The nine-month intervention wave will be mentored by INS study personnel who will accompany and support district MOH supervisors as they implement at the facility level. Over the first week of each iterative cycle, facility teams populate and interpret the HCAT, develop process maps, define one to two micro-interventions and indicators to monitor these modifications. Facility teams receive two mentorship visits by district supervisors and study personnel for the first month, followed by monthly visits throughout intensive implementation.
  Sustainment phase (depending on implementation wave allocation): district supervisors will independently lead implementation, with financial support for travel to clinics and to hold meetings, but without intensive support from study personnel.
  Arms: intervention health facilities

SUMMARY:
Undiagnosed and untreated hypertension is a main driver of cardiovascular disease, affecting disproportionately low and middle-income countries, where guidelines to screen and manage hypertension are poorly used. More than 13% of Mozambique adults are infected with HIV, and over 900,000 are on anti-retroviral therapy. HIV clinics are the only services within primary care providing continued care, and can be used to standardize and scale the hypertension care cascade. Hypertension affects 40% of Mozambican adults, and thus HIV and HTN often coexist in the same person.

The investigators propose to use low-cost tools that improve service performance, promote routine hypertension diagnosis and management, and ameliorate flow through the hypertension cascade, thus improving patients outcomes. Building on a current project some districts of two provinces of central Mozambique, the investigators will establish scientific evidence on the effectiveness of a tool that uses cycles of evaluation and improvement of health system, to address the hypertension care cascade in HIV-infected people. The investigators will strengthen the framework currently in use (based on nurses) setting a novel modality delivered by district health supervisors, and will expand the geographic study area by adding 6 districts of one additional province in southern Mozambique (Maputo Province), to create a foundation for national scale-up.

The Project planning phase (two years) will develop a multi-sectoral partnership of key stakeholders, establish national technical working groups with the participation of the provinces, and identify key facilitators and barriers that could affect uptake of the results, integration of high blood pressure and HIV services, scale-up to the entire country, and sustainability of the tested framework. Additionally, the investigators will i) conduct a six-months pilot study to assess feasibility and acceptability of the district supervisor-led intervention in one primary care facility; and, ii) redesign tools and standard operating procedures, as necessary. During the implementation phase (last three years) the investigators will deploy the district-based dissemination and implementation randomized trial in 18 health facilities - using an intervention that involves assessment, effectiveness evaluation, promotion of local uptake, implementation and maintenance - and determine the costs of the hypertension care cascade optimization, by estimating the total incremental costs.

DETAILED DESCRIPTION:
In Mozambique HIV prevalence is over 13% and hypertension (HTN) affects 40% of adults. HIV and HTN comorbidity is increasing with the aging of HIV-infected population and expansion of antiretroviral therapy (ART), but guideline application for HTN screening and management remains low and uneven. Around 14% of adults are aware of their HTN status and only 3% of those with HTN have their condition controlled. The HIV treatment platform is the only broadly implemented chronic care service and provides an opportunity to standardize and scale HTN screening and management.

Systems-level implementation strategies may reduce drop-offs along the HTN cascade, improve service quality, and maximize availability of efficacious HTN medicines. Systems engineering tools can identify drivers of inefficiency, support locally informed provider decision-making to prioritize solutions, and improve integration of services to reduce inefficiencies in complex, multi-step health services using simple, low cost, iterative adaptations in service delivery design. The participation of frontline staff and senior management champions in this process improves patient outcomes.

The investigators aim to describe HTN care cascade at the health facility level and use it as the entry point for systems optimization of HIV services, using cascade analysis and associated systems engineering tools. In central Mozambique a Systems Analysis and Improvement Approach (SAIA) identified HTN cascade steps for PLHIV, developed a HTN Cascade Analysis Tool (HCAT), mapped data sources, and developed a registry to populate the HCAT and capture study outcomes from outpatient registries and patient charts (SAIA-HTN). Building on this, our project will 'scale out' through the novel modality of delivery by district health supervisors, and 'scale up' by expanding to six districts in one additional province (SCALE SAIA-HTN). It also aims at developing a dissemination and implementation model to serve as a foundation for national scaling.

Projects Aims:

1. To develop a multi-sectoral partnership of key stakeholders and establish HTN technical working groups at the national level and participating provinces;
2. To identify key facilitators and barriers that could affect the adoption, integration, scale-up and sustainment of the SAIA-HTN implementation strategy;
3. To conduct a pilot study to assess feasibility and acceptability of the district MOH supervisor-led SAIA-HTN intervention over six months in one primary care facility (to redesign tools and standard operating procedures as necessary);
4. Develop a district-based dissemination and implementation of SAIA-HTN (SCALE SAIA-HTN) using the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) model to evaluate the program: a. Determine the proportion of health facilities and population in the six districts reached, and identification of sub-groups not reached (target: 33% of facilities and 80% HIV+ adults reached); b.Assess the intervention effect on HTN process measures (BP screening, HTN diagnosis, HTN medication initiation, maintenance on HTN treatment), and HTN treatment effectiveness (HTN control, HIV viral load suppression); c.Determine the proportion of districts and facilities adopting the intervention (target: 95%), and explore the determinants of adoption identified using the Organizational Readiness for Implementing Change (ORIC); d.Determine core elements of the scaled SAIA-HTN implementation process and describe drivers of success/failure using the Consolidated Framework for Implementation Research (CFIR); e.Calculate the proportion of districts sustaining the intervention 9, 18, 27 months post-introduction (target: >90% at 9 months, >80% at 18 months, and >65% at 27 months).
5. Determine the costs of SCALE SAIA-HTN for care cascade optimization, including total incremental and unit costs of integrating HTN diagnosis and management into HIV care.

Methods: The investigators will use the SAIA strategy to visualize and quantify interconnected service delivery steps, informed by previous SAIA research, epidemiologic research on HTN, and ongoing SAIA-HTN research to optimize HTN screening, care and treatment for PLHIV in central Mozambique (to evaluate SAIA-HTN's effectiveness on systems' and patient-level health outcomes for PLHIV).

Study Plan: The investigators will use multiple novel implementation science methods to understand and explain what influences implementation outcomes, including i) the CFIR to identify barriers and facilitators (determinants) to implementation, ii) the ORIC scale to assesses readiness for change as an organizational-level determinant of adoption, and iii) the RE-AIM evaluative Framework, which measures the active ingredients for public health impact (Reach, Effectiveness, Adoption, Implementation and Maintenance).

Planning phase: The investigators will mobilize a multi-sectoral stakeholder partnership, conduct a needs assessment (to evaluate facilitators and barriers that could affect adoption, integration, scale-up and sustainment of SCALE SAIA-HTN in the two provinces), and pilot the intervention's feasibility and acceptability over six months in one clinics (to refine implementation procedures for follow-on scaling out and scaling up).Implementation phase: 'scale out' SAIA-HTN to test a novel delivery modality (using district supervisors), 'scale up' to cover six districts in Maputo province, and evaluate its impact on cascade performance and patient outcomes. The investigators will randomly allocate health facilities from the six districts in Maputo Province into three implementation waves, staggered by nine months (27 months total).

The SAIA-HTN implementation strategy uses an iterative, five-step process applied at the facility level to give clinic staff and managers a systems view of cascade performance, identify priority areas for improvement, discern modifiable solutions, and test workflow modifications.

SCALE SAIA-HTN will test integration and scale up of SAIA-HTN through routine management systems relying on district Ministry of Health (MOH) supervisors as the disseminating agents (rather than research nurses), in three facilities per district during a nine-month intensive phase (mentored by study assistants), and subsequent sustainment phase (led independently by district MOH supervisors). Based on trial results, the investigators will model out the costs and potential benefits on HTN management for PLHIV given different scale-up scenarios nationwide. The trial will culminate in the development and dissemination of the SCALE SAIA-HTN package, summarizing trial results and providing implementation and cost guidance to inform policy development and support national scale-up through routine management structures.

Study design: phased-in (stepped wedge) with random assignment of two districts to each of the three nine-month intervention waves, to reach six districts in Maputo Province by the end of the trial.

Study Setting: Maputo Province (population of >1.5 million inhabitants; >98% of formal health services offered through public sector clinics). Health facilities with highest numbers of active HIV+ patients on ART will be enrolled.

Study Team: This project brings together a diverse and uniquely qualified team of cardiovascular, HIV, community surveys, health systems, and implementation scientists.

Procedures Stakeholders meetings: to create a multi-sectoral partnership of key stakeholders and establish HTN technical working groups (TWG) at the national level and with participating provinces.

Stakeholder field visits to SAIA-HTN trial in central Mozambique: for key personnel and district MOH supervisors from the pilot facility.

Orientation meetings/workshops: for introducing SCALE SAIA-HTN, the implementation approach, and evaluation design to study investigators, provincial MOH managers, and district MOH supervisors in each province, who will review and agree on study procedures, and clinical and organizational skills-building approaches. Throughout the two phases of the project the TWG will inform on mediators and mechanisms of action, scale-up and sustainment efforts, and ensure responsiveness to local needs; at end of the planning phase, the TWG will review findings, discuss necessary adaptations and refine SCALE SAIA-HTN for the implementation phase.

Standardized readiness assessments: in the six first wave health facilities to assess structural and organizational readiness to deliver HTN services (ORIC measures, staffing levels, attributes and training, availability of essential commodities, equipment and supplies, and infrastructure) and repeated for subsequent waves prior to launching intensive implementation phases.

Pilot study: Outpatient staff managing HIV/CVD care and district MOH supervisors will participate in orientation training for the feasibility and acceptability of the SCALE SAIA-HTN intervention, which will be carried out over six months in one primary care facility. Tools and standard operating procedures will be redesigned as necessary for the implementation phase. Facility-based HTN screening will be carried out by nurses at entry into the pilot facility; all hypertensive (new and existing) patients will be recruited, with the support of district supervisors and study teams. Feasibility and acceptability will include i) measurement of intervention fidelity, reach and exposure, and adoption; ii) knowledge and competency questionnaire to health personnel. Follow-up visits to both monitor and support implementation will be carried out twice in the first month, and monthly thereafter. Additional data will be collected by: focus group discussion (FGD) with key staff to assess acceptability of content and delivery of the intervention; questionnaire to participating staff pre and post-intervention; key informant interviews with the district supervisors, facility managers and frontline staff.

Evaluate programs' Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) Reach: determine the number, proportion/representativeness of individuals reached by interventions; use study reports to estimate the proportion of facilities in the six districts reached by SCALE SAIA-HTN (target: 30%); determine the number and proportion of HIV-infected adults with HTN reached (target: 80%).

Effectiveness: HTN treatment effectiveness (primary effectiveness outcome: HTN control, Secondary outcomes: HIV viral load suppression, proportion of HIV- infected patients screened for HTN in outpatient services, HTN diagnosis, HTN prescription of eligible patients, >90% patient adherence to HTN treatment).

Adoption: ORIC assessment scale (target of 95%) used to six frontline staff working across the HIV-HTN cascade and facility leadership in each clinic (n=108), and two supervisors (NCD and HIV) from each district (n=12) to describe determinants of adoption.

Implementation: Tools at CFIR website will be adapted to gather data via interviews and FGDs with facility and district staff (qualitative), intervention meeting minutes (qualitative), and annual quantitative questionnaires to quantify facility structural determinants of implementation of HTN management guidelines.

Maintenance. Proportion of districts sustaining the intervention as designed 9, 18 and 27 months post-introduction (target: >90% at 9 months, >80% at 18 months, and >65% at 27 months). In-depth interviews and FGDs to probe district/facility perspectives on determinants of sustainment

Determination of the costs of SCALE SAIA-HTN for care cascade optimization: total incremental and unit costs of integrating HTN diagnosis and management into HIV care. For cost estimation activity-based cost menus will identify start up and recurrent activities, and measure resource use and costs from design through implementation. Cost metrics will include the total incremental costs and average unit costs.

ELIGIBILITY:
Inclusion Criteria:

* Primary care facility with ongoing cohort of ART patients (minimum 800 patients)

Exclusion Criteria:

* Health facility unaccessible during part of the year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
REACH Year 3 - health facilities | Year 3
  Proportion of health facilities in Maputo Province reached and identification of sub-groups not reached (target: 33% of facilities and 80% HIV+ adults reached).
REACH Year 3 - population | Year 3
  Proportion of population in Maputo Province reached and identification of sub-groups not reached (target: 33% of facilities and 80% HIV+ adults reached).
REACH Year 4 - health facilities | Year 4
  Proportion of health facilities in Maputo Province reached and identification of sub-groups not reached (target: 33% of facilities and 80% HIV+ adults reached).
REACH Year 4 - population | Year 4
  Proportion of population in Maputo Province reached and identification of sub-groups not reached (target: 33% of facilities and 80% HIV+ adults reached).
REACH Year 5 - health facilities | Year 5
  Proportion of health facilities in Maputo Province reached and identification of sub-groups not reached (target: 33% of facilities and 80% HIV+ adults reached).
REACH Year 5 - population | Year 5
  Proportion of population in Maputo Province reached and identification of sub-groups not reached (target: 33% of facilities and 80% HIV+ adults reached).
Screening EFFECTIVENESS Year 3 - BP screening coverage | Year 3
  Proportion of adult patients screened
Screening EFFECTIVENESS Year 3 - Prevalence | Year 3
  Prevalence of HTN among those screened
Screening EFFECTIVENESS Year 3 - Proportion initiating HTN medication | Year 3
  Proportion initiating HTN medication
Screening EFFECTIVENESS Year 3 - Proportion maintained on treatment | Year 3
  Proportion maintained on treatment
Screening EFFECTIVENESS Year 4 - BP screening coverage | Year 4
  Proportion of adult patients screened
Screening EFFECTIVENESS Year 4 - Prevalence of HTN among those screened | Year 4
  Prevalence of HTN among those screened
Screening EFFECTIVENESS Year 4 - Proportion initiating HTN medication | Year 4
  Proportion initiating HTN medication
Screening EFFECTIVENESS Year 4 - Proportion maintained on treatment | Year 4
  Proportion maintained on treatment
Screening EFFECTIVENESS Year 5 - BP screening coverage | Year 5
  Proportion of adult patients screened
Screening EFFECTIVENESS Year 5 - Prevalence of HTN among those screened | Year 5
  Prevalence of HTN among those screened
Screening EFFECTIVENESS Year 5 - Proportion initiating HTN medication | Year 5
  Proportion initiating HTN medication
Screening EFFECTIVENESS Year 5 - Proportion maintained on treatment | Year 5
  Proportion maintained on treatment
Treatment EFFECTIVENESS Year 3 - HTN control | Year 3
  proportion of patients with HTN controlled
Treatment EFFECTIVENESS Year 3 - HIV viral load suppression | Year 3
  proportion of HIV patients with viral load suppression
Treatment EFFECTIVENESS Year 4 - HTN control | Year 4
  proportion of patients with HTN controlled
Treatment EFFECTIVENESS Year 4 - HIV viral load suppression | Year 4
  proportion of HIV patients with viral load suppression
Treatment EFFECTIVENESS Year 5 - HTN control | Year 5
  proportion of patients with HTN controlled
Treatment EFFECTIVENESS Year 5 - HIV viral load suppression | Year 5
  proportion of HIV patients with viral load suppression
ADOPTION Year 4 - districts and facilities | Year 4
  Proportion of districts and facilities adopting the intervention (target: 95%)
ADOPTION Year 4 - Organizational Readiness for Implementing Change (ORIC) | Year 4
  Assess the extent to which organizational members are psychologically and behaviorally prepared to implement change (change commitment and change efficacy) using the Likert scale from 1("disagree") to 5 ("strongly agree")
ADOPTION Year 5 - districts and facilities | Year 5
  Proportion of districts and facilities adopting the intervention (target: 95%)
ADOPTION Year 5 - Organizational Readiness for Implementing Change (ORIC) | Year 5
  Assess the extent to which organizational members are psychologically and behaviorally prepared to implement change (change commitment and change efficacy) using the Likert scale from 1("disagree") to 5 ("strongly agree")
IMPLEMENTATION Year 3 - Determine core elements of the scaled SAIA-HTN implementation process | Year 3
  Use the Consolidated Framework for Implementation Research to guide examination of implementation process through semi-structured in-depth interviews and focus group discussions
IMPLEMENTATION Year 3 - drivers of success/failure | Year 3
  Use the Consolidated Framework for Implementation Research (CFIR) to describe determinants of success and failure found across implementing districts and facilities through semi-structured in-depth interviews and focus group discussions
IMPLEMENTATION Year 4 - Determine core elements of the scaled SAIA-HTN implementation process | Year 4
  Use the Consolidated Framework for Implementation Research to guide examination of implementation process through semi-structured in-depth interviews and focus group discussions
IMPLEMENTATION Year 4 - drivers of success/failure | Year 4
  Use the Consolidated Framework for Implementation Research (CFIR) to describe determinants of success and failure found across implementing districts and facilities through semi-structured in-depth interviews and focus group discussions
IMPLEMENTATION Year 5 - Determine core elements of the scaled SAIA-HTN implementation process | Year 5
  Use the Consolidated Framework for Implementation Research to guide examination of implementation process through semi-structured in-depth interviews and focus group discussions
IMPLEMENTATION Year 5 - drivers of success/failure | Year 5
  Use the Consolidated Framework for Implementation Research (CFIR) to describe determinants of success and failure found across implementing districts and facilities through semi-structured in-depth interviews and focus group discussions
MAINTENANCE Year 3 | Year 3
  Proportion of districts sustaining the intervention as designed 9 months post introduction (first wave of health facilities)
MAINTENANCE Year 4 | Year 4
  Proportion of districts sustaining the intervention as designed 18 and 27 months post introduction for second and first wave of health facilities, respectively
MAINTENANCE Year 5 | Year 5
  Proportion of districts sustaining the intervention as designed 9, 18 and 27 months post introduction for third, second and first wave of health facilities, respectively
COST ESTIMATION Year 4 | Year 4
  estimate its incremental costs of SCALE SAIA HTN compared to the status quo
COST ESTIMATION Year 5 | Year 5
  Estimate incremental costs of SCALE SAIA HTN compared to the status quo
ESTIMATING AFFORDABILITY AND BUDGET IMPACT Year 4 | Year 4
  Estimate the cost per person screened and treated for HTN
ESTIMATING AFFORDABILITY AND BUDGET IMPACT Year 5 | Year5
  Estimate the cost per person screened and treated for HTN
ECONOMIC EVALUATION Year 4 | Year 4
  Comparing the total costs of HTN diagnosis and care as a proportion of the HIV care budget and estimate QALYs
ECONOMIC EVALUATION Year 5 | Year 5
  Comparing the total costs of HTN diagnosis and care as a proportion of the HIV care budget and estimate QALYs

CONTACTS AND LOCATIONS:
Overall Officials: Ana OH Mocumbi, MD PhD, Principal Investigator — Eduardo Mondlane University
Locations (6):
- Mozambique (6):
  - Centro de Saude da Ponta do Ouro, Bela Vista, Maputo Province
  - Centro de Saude de Matutuine, Bela Vista, Maputo Province
  - Centro de Saude de Salamanga, Bela Vista, Maputo Province
  - Centro de Saúde de Magude, Magude, Maputo Province
  - Centro de Saúde de Motaze, Magude, Maputo Province
  - Centro de Saúde de Chichuco, Magude

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Burden of Metabolic Risk Factors for Chronic Diseases Collaboration. Cardiovascular disease, chronic kidney disease, and diabetes mortality burden of cardiometabolic risk factors from 1980 to 2010: a comparative risk assessment. Lancet Diabetes Endocrinol. 2014 Aug;2(8):634-47. doi: 10.1016/S2213-8587(14)70102-0. Epub 2014 May 16. PMID 24842598
- [Background] Kengne AP, Ntyintyane LM, Mayosi BM. A systematic overview of prospective cohort studies of cardiovascular disease in sub-Saharan Africa. Cardiovasc J Afr. 2012 Mar;23(2):103-12. doi: 10.5830/CVJA-2011-042. Epub 2011 Sep 7. PMID 21901226
- [Background] Ibrahim MM, Damasceno A. Hypertension in developing countries. Lancet. 2012 Aug 11;380(9841):611-9. doi: 10.1016/S0140-6736(12)60861-7. PMID 22883510
- [Background] van de Vijver S, Akinyi H, Oti S, Olajide A, Agyemang C, Aboderin I, Kyobutungi C. Status report on hypertension in Africa--consultative review for the 6th Session of the African Union Conference of Ministers of Health on NCD's. Pan Afr Med J. 2013 Oct 5;16:38. doi: 10.11604/pamj.2013.16.38.3100. eCollection 2013. PMID 24570798
- [Background] Ministerio da Saude. Relatorio Anual 2017 HIV. Maputo, Mocambique: Ministerio da Saude; 2014.
- [Background] Jessen N, Damasceno A, Silva-Matos C, Tuzine E, Madede T, Mahoque R, Padrao P, Mbofana F, Polonia J, Lunet N. Hypertension in Mozambique: trends between 2005 and 2015. J Hypertens. 2018 Apr;36(4):779-784. doi: 10.1097/HJH.0000000000001618. PMID 29210894
- [Background] Antonello VS, Antonello IC, Grossmann TK, Tovo CV, Pupo BB, Winckler Lde Q. Hypertension--an emerging cardiovascular risk factor in HIV infection. J Am Soc Hypertens. 2015 May;9(5):403-7. doi: 10.1016/j.jash.2015.03.008. Epub 2015 Mar 28. PMID 25979413
- [Background] Lloyd-Sherlock P, Ebrahim S, Grosskurth H. Is hypertension the new HIV epidemic? Int J Epidemiol. 2014 Feb;43(1):8-10. doi: 10.1093/ije/dyu019. Epub 2014 Feb 3. No abstract available. PMID 24491955
- [Background] Medina-Torne S, Ganesan A, Barahona I, Crum-Cianflone NF. Hypertension is common among HIV-infected persons, but not associated with HAART. J Int Assoc Physicians AIDS Care (Chic). 2012 Jan-Feb;11(1):20-5. doi: 10.1177/1545109711418361. Epub 2011 Aug 29. PMID 21876213
- [Background] Schouten J, Wit FW, Stolte IG, Kootstra NA, van der Valk M, Geerlings SE, Prins M, Reiss P; AGEhIV Cohort Study Group. Cross-sectional comparison of the prevalence of age-associated comorbidities and their risk factors between HIV-infected and uninfected individuals: the AGEhIV cohort study. Clin Infect Dis. 2014 Dec 15;59(12):1787-97. doi: 10.1093/cid/ciu701. Epub 2014 Sep 2. PMID 25182245
- [Background] Marcus JL, Chao CR, Leyden WA, Xu L, Quesenberry CP Jr, Klein DB, Towner WJ, Horberg MA, Silverberg MJ. Narrowing the Gap in Life Expectancy Between HIV-Infected and HIV-Uninfected Individuals With Access to Care. J Acquir Immune Defic Syndr. 2016 Sep 1;73(1):39-46. doi: 10.1097/QAI.0000000000001014. PMID 27028501
- [Background] Dzudie A, Rayner B, Ojji D, Schutte AE, Twagirumukiza M, Damasceno A, Ba SA, Kane A, Kramoh E, Anzouan Kacou JB, Onwubere B, Cornick R, Sliwa K, Anisiuba B, Mocumbi AO, Ogola E, Awad M, Nel G, Otieno H, Toure AI, Kingue S, Kengne AP, Perel P, Adler A, Poulter N, Mayosi B; PASCAR Task Force on Hypertension. Roadmap to Achieve 25% Hypertension Control in Africa by 2025. Glob Heart. 2018 Mar;13(1):45-59. doi: 10.1016/j.gheart.2017.06.001. Epub 2017 Oct 16. PMID 29042191
- [Background] Kayima J, Wanyenze RK, Katamba A, Leontsini E, Nuwaha F. Hypertension awareness, treatment and control in Africa: a systematic review. BMC Cardiovasc Disord. 2013 Aug 2;13:54. doi: 10.1186/1471-2261-13-54. PMID 23915151
- [Background] Baekken M, Os I, Sandvik L, Oektedalen O. Hypertension in an urban HIV-positive population compared with the general population: influence of combination antiretroviral therapy. J Hypertens. 2008 Nov;26(11):2126-33. doi: 10.1097/HJH.0b013e32830ef5fb. PMID 18854751
- [Background] Sherer R, Solomon S, Schechter M, Nachega JB, Rockstroh J, Zuniga JM. HIV provider-patient communication regarding cardiovascular risk: results from the AIDS Treatment for Life International Survey. J Int Assoc Provid AIDS Care. 2014 Jul-Aug;13(4):342-5. PMID 25513031
- [Background] Lichtenstein KA, Armon C, Buchacz K, Chmiel JS, Buckner K, Tedaldi E, Wood K, Holmberg SD, Brooks JT; HOPS Investigators. Provider compliance with guidelines for management of cardiovascular risk in HIV-infected patients. Prev Chronic Dis. 2013;10:E10. doi: 10.5888/pcd10.120083. PMID 23347705
- [Background] Ameh S, Klipstein-Grobusch K, Musenge E, Kahn K, Tollman S, Gomez-Olive FX. Effectiveness of an Integrated Approach to HIV and Hypertension Care in Rural South Africa: Controlled Interrupted Time-Series Analysis. J Acquir Immune Defic Syndr. 2017 Aug 1;75(4):472-479. doi: 10.1097/QAI.0000000000001437. PMID 28640065
- [Background] Rabkin M, Kruk ME, El-Sadr WM. HIV, aging and continuity care: strengthening health systems to support services for noncommunicable diseases in low-income countries. AIDS. 2012 Jul 31;26 Suppl 1:S77-83. doi: 10.1097/QAD.0b013e3283558430. PMID 22781180
- [Background] Wagner AD, Gimbel S, Asbjornsdottir KH, Cherutich P, Coutinho J, Crocker J, Cruz E, Cuembelo F, Cumbe V, Eastment M, Einberg J, Floriano F, Gaitho D, Guthrie BL, John-Stewart G, Kral AH, Lambdin BH, Liu S, Maina M, Manaca N, Matsuzaki M, Mattox L, Mburu N, McClelland RS, Micek MA, Mocumbi AO, Muanido A, Nduati R, Njuguna IN, Oluoch G, Oyiengo LB, Ronen K, Soi C, Wagenaar BH, Wanje G, Wenger LD, Sherr K. Cascade Analysis: An Adaptable Implementation Strategy Across HIV and Non-HIV Delivery Platforms. J Acquir Immune Defic Syndr. 2019 Dec;82 Suppl 3(Suppl 3):S322-S331. doi: 10.1097/QAI.0000000000002220. PMID 31764270
- [Background] Kwarisiima D, Atukunda M, Owaraganise A, Chamie G, Clark T, Kabami J, Jain V, Byonanebye D, Mwangwa F, Balzer LB, Charlebois E, Kamya MR, Petersen M, Havlir DV, Brown LB. Hypertension control in integrated HIV and chronic disease clinics in Uganda in the SEARCH study. BMC Public Health. 2019 May 6;19(1):511. doi: 10.1186/s12889-019-6838-6. PMID 31060545
- [Background] Ngu RC, Choukem SP, Dimala CA, Ngu JN, Monekosso GL. Prevalence and determinants of selected cardio-metabolic risk factors among people living with HIV/AIDS and receiving care in the South West Regional Hospitals of Cameroon: a cross-sectional study. BMC Res Notes. 2018 May 16;11(1):305. doi: 10.1186/s13104-018-3444-0. PMID 29769110
- [Background] van Heerden A, Barnabas RV, Norris SA, Micklesfield LK, van Rooyen H, Celum C. High prevalence of HIV and non-communicable disease (NCD) risk factors in rural KwaZulu-Natal, South Africa. J Int AIDS Soc. 2017 Oct;20(2):e25012. doi: 10.1002/jia2.25012. PMID 29064168
- [Background] Muddu M, Tusubira AK, Sharma SK, Akiteng AR, Ssinabulya I, Schwartz JI. Integrated Hypertension and HIV Care Cascades in an HIV Treatment Program in Eastern Uganda: A Retrospective Cohort Study. J Acquir Immune Defic Syndr. 2019 Aug 15;81(5):552-561. doi: 10.1097/QAI.0000000000002067. PMID 31045649
- [Background] Womak J, Byrne A, Flume O, Kaplan G, Toussaint J. Going lean in health care: Available online at: www.ihi.org; 2005.
- [Background] Weinberg M, Fuentes JM, Ruiz AI, Lozano FW, Angel E, Gaitan H, Goethe B, Parra S, Hellerstein S, Ross-Degnan D, Goldmann DA, Huskins WC. Reducing infections among women undergoing cesarean section in Colombia by means of continuous quality improvement methods. Arch Intern Med. 2001 Oct 22;161(19):2357-65. doi: 10.1001/archinte.161.19.2357. PMID 11606152
- [Background] Aarons GA, Sklar M, Mustanski B, Benbow N, Brown CH. "Scaling-out" evidence-based interventions to new populations or new health care delivery systems. Implement Sci. 2017 Sep 6;12(1):111. doi: 10.1186/s13012-017-0640-6. PMID 28877746
- [Background] Gimbel S, Mocumbi AO, Asbjornsdottir K, Coutinho J, Andela L, Cebola B, Craine H, Crocker J, Hicks L, Holte S, Hossieke R, Itai E, Levin C, Manaca N, Murgorgo F, Nhumba M, Pfeiffer J, Ramiro I, Ronen K, Sotoodehnia N, Uetela O, Wagner A, Weiner BJ, Sherr K. Systems analysis and improvement approach to optimize the hypertension diagnosis and care cascade for PLHIV individuals (SAIA-HTN): a hybrid type III cluster randomized trial. Implement Sci. 2020 Mar 6;15(1):15. doi: 10.1186/s13012-020-0973-4. PMID 32143657
- [Background] Nelson E, Batalden P, Godfrey M. Quality by Design: A Clinical microsystems Approach. San Francisco: Jossey-Bass; 2007.
- [Background] Curry LA, Spatz E, Cherlin E, Thompson JW, Berg D, Ting HH, Decker C, Krumholz HM, Bradley EH. What distinguishes top-performing hospitals in acute myocardial infarction mortality rates? A qualitative study. Ann Intern Med. 2011 Mar 15;154(6):384-90. doi: 10.7326/0003-4819-154-6-201103150-00003. PMID 21403074
- [Background] Sherr K, Gimbel S, Rustagi A, Nduati R, Cuembelo F, Farquhar C, Wasserheit J, Gloyd S; With input from the SAIA Study Team. Systems analysis and improvement to optimize pMTCT (SAIA): a cluster randomized trial. Implement Sci. 2014 May 8;9:55. doi: 10.1186/1748-5908-9-55. PMID 24885976
- [Background] Rustagi AS, Gimbel S, Nduati R, Cuembelo Mde F, Wasserheit JN, Farquhar C, Gloyd S, Sherr K; with input from the SAIA Study Team. Implementation and Operational Research: Impact of a Systems Engineering Intervention on PMTCT Service Delivery in Cote d'Ivoire, Kenya, Mozambique: A Cluster Randomized Trial. J Acquir Immune Defic Syndr. 2016 Jul 1;72(3):e68-76. doi: 10.1097/QAI.0000000000001023. PMID 27082507
- [Background] Gimbel S, Rustagi AS, Robinson J, Kouyate S, Coutinho J, Nduati R, Pfeiffer J, Gloyd S, Sherr K, Granato SA, Kone A, Cruz E, Manuel JL, Zucule J, Napua M, Mbatia G, Wariua G, Maina M; with input from the SAIA study team. Evaluation of a Systems Analysis and Improvement Approach to Optimize Prevention of Mother-To-Child Transmission of HIV Using the Consolidated Framework for Implementation Research. J Acquir Immune Defic Syndr. 2016 Aug 1;72 Suppl 2(Suppl 2):S108-16. doi: 10.1097/QAI.0000000000001055. PMID 27355497
- [Background] Wozniak G, Khan T, Gillespie C, Sifuentes L, Hasan O, Ritchey M, Kmetik K, Wynia M. Hypertension Control Cascade: A Framework to Improve Hypertension Awareness, Treatment, and Control. J Clin Hypertens (Greenwich). 2016 Mar;18(3):232-9. doi: 10.1111/jch.12654. Epub 2015 Sep 4. PMID 26337797
- [Background] Berry KM, Parker WA, Mchiza ZJ, Sewpaul R, Labadarios D, Rosen S, Stokes A. Quantifying unmet need for hypertension care in South Africa through a care cascade: evidence from the SANHANES, 2011-2012. BMJ Glob Health. 2017 Aug 16;2(3):e000348. doi: 10.1136/bmjgh-2017-000348. eCollection 2017. PMID 29082013
- [Background] Nilsen P. Making sense of implementation theories, models and frameworks. Implement Sci. 2015 Apr 21;10:53. doi: 10.1186/s13012-015-0242-0. PMID 25895742
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Weiner BJ. A theory of organizational readiness for change. Implement Sci. 2009 Oct 19;4:67. doi: 10.1186/1748-5908-4-67. PMID 19840381
- [Background] Shea CM, Jacobs SR, Esserman DA, Bruce K, Weiner BJ. Organizational readiness for implementing change: a psychometric assessment of a new measure. Implement Sci. 2014 Jan 10;9:7. doi: 10.1186/1748-5908-9-7. PMID 24410955
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Damasceno A, Azevedo A, Silva-Matos C, Prista A, Diogo D, Lunet N. Hypertension prevalence, awareness, treatment, and control in mozambique: urban/rural gap during epidemiological transition. Hypertension. 2009 Jul;54(1):77-83. doi: 10.1161/HYPERTENSIONAHA.109.132423. Epub 2009 May 26. PMID 19470872
- [Background] Wagenaar BH, Gimbel S, Hoek R, Pfeiffer J, Michel C, Manuel JL, Cuembelo F, Quembo T, Afonso P, Gloyd S, Sherr K. Stock-outs of essential health products in Mozambique - longitudinal analyses from 2011 to 2013. Trop Med Int Health. 2014 Jul;19(7):791-801. doi: 10.1111/tmi.12314. Epub 2014 Apr 11. PMID 24724617
- [Background] Sherr K, Cuembelo F, Michel C, Gimbel S, Micek M, Kariaganis M, Pio A, Manuel JL, Pfeiffer J, Gloyd S. Strengthening integrated primary health care in Sofala, Mozambique. BMC Health Serv Res. 2013;13 Suppl 2(Suppl 2):S4. doi: 10.1186/1472-6963-13-S2-S4. Epub 2013 May 31. PMID 23819552
- [Background] National Statistic Institute. Mozambique Demographich Health Survey Final Report, 2011. Maputo, Mozambique; 2012. 2012.
- [Background] Manafe N, Matimbe RN, Daniel J, Lecour S, Sliwa K, Mocumbi AO. Hypertension in a resource-limited setting: Poor Outcomes on Short-term Follow-up in an Urban Hospital in Maputo, Mozambique. J Clin Hypertens (Greenwich). 2019 Dec;21(12):1831-1840. doi: 10.1111/jch.13732. Epub 2019 Nov 25. PMID 31769184
- [Background] Mocumbi AO, Ferreira MB, Sidi D, Yacoub MH. A population study of endomyocardial fibrosis in a rural area of Mozambique. N Engl J Med. 2008 Jul 3;359(1):43-9. doi: 10.1056/NEJMoa0708629. PMID 18596273
- [Background] Mocumbi AO, Langa DC, Chicumbe S, Schumacher AE, Al-Delaimy WK. Incorporating selected non-communicable diseases into facility-based surveillance systems from a resource-limited setting in Africa. BMC Public Health. 2019 Feb 4;19(1):147. doi: 10.1186/s12889-019-6473-2. PMID 30717732
- [Background] Klein K, Dansereau F, Hall R. Levels issues in theory development, data collection and analysis. Academy of Management Review 1994;19:195-229.
- [Background] Klein K, Kozlowski S. From micro to meso: critical steps in conceptualizing and conducting multilevel research. Organizational Research Methods 2000;3:211-36.
- [Background] LeBreton J, James L, Lindell M. Recent issues regarding r(WG), r*(WG), r(WG)(J), and r*(WG)(J). Organizational Research Methods 2005;8:128-38.
- [Background] LeBreton J, Senter J. Answers to 20 questions about interrater reliability and interrater agreement. Organizational Research Methods 2008;11:815-52.
- [Background] Krueger R, Casey MA. Focus groups: a practical guide for applied research: Sage Publications, Thousand Oaks, CA. ; 2000.
- [Background] Strauss A, Corbin J. Basics of qualitative research: Techniques and procedures for developing grounded theory. Thousand Oaks, California: SAGE Publications; 1998.
- [Background] Choosing Interventions that are Cost-Effective. Estimates of Unit Costs of Patient Services. World Health Organization. (Accessed September 29, 2016, at http://www.who.int/choice/cost-effectiveness/inputs/health_service/en/.)
- [Background] Bilinski A, Neumann P, Cohen J, Thorat T, McDaniel K, Salomon JA. When cost-effective interventions are unaffordable: Integrating cost-effectiveness and budget impact in priority setting for global health programs. PLoS Med. 2017 Oct 2;14(10):e1002397. doi: 10.1371/journal.pmed.1002397. eCollection 2017 Oct. PMID 28968399
- [Background] Sanders GD, Neumann PJ, Basu A, Brock DW, Feeny D, Krahn M, Kuntz KM, Meltzer DO, Owens DK, Prosser LA, Salomon JA, Sculpher MJ, Trikalinos TA, Russell LB, Siegel JE, Ganiats TG. Recommendations for Conduct, Methodological Practices, and Reporting of Cost-effectiveness Analyses: Second Panel on Cost-Effectiveness in Health and Medicine. JAMA. 2016 Sep 13;316(10):1093-103. doi: 10.1001/jama.2016.12195. PMID 27623463
- [Background] Finch AP, Brazier JE, Mukuria C. What is the evidence for the performance of generic preference-based measures? A systematic overview of reviews. Eur J Health Econ. 2018 May;19(4):557-570. doi: 10.1007/s10198-017-0902-x. Epub 2017 May 30. PMID 28560520
- [Derived] Hazim CE, Dobe I, Pope S, Asbjornsdottir KH, Augusto O, Bruno FP, Chicumbe S, Lumbandali N, Mate I, Ofumhan E, Patel S, Rafik R, Sherr K, Tonwe V, Uetela O, Watkins D, Gimbel S, Mocumbi AO. Scaling-up and scaling-out the Systems Analysis and Improvement Approach to optimize the hypertension diagnosis and care cascade for HIV infected individuals (SCALE SAIA-HTN): a stepped-wedge cluster randomized trial. Implement Sci Commun. 2024 Mar 20;5(1):27. doi: 10.1186/s43058-024-00564-1. PMID 38509605